CLINICAL TRIAL: NCT03775928
Title: Phase Ⅱ Study of Compare Apatinib Plus Capecitabine Versus Capecitabine in Maintenance Therapy for Patients With Advanced Triple-negative Breast Cancer
Brief Title: Compare Apatinib Plus Capecitabine Versus Capecitabine in Maintenance Therapy for Patients With Advanced Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, clinical professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — apatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib + Capecitabine (Experimental): Apatinib 425mg d1-21+ capecitabine 1000mg/m2 bid d1-14, q21d
  Interventions: Drug: Apatinib; Drug: capecitabine
- Capecitabine (Active Comparator): capecitabine 1000mg/m2 bid d1-14, q21d
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Apatinib — apatinib 425mg qd po
  Arms: Apatinib + Capecitabine
Drug: capecitabine — capecitabine 1000mg/m2 bid d1-d14

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive apatinib plus capecitabine or capecitabine for maintenance therapy of patients with with advanced triple-negative breast cancer

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) has the characteristics of early onset, high malignancy, less treatment, and resistance to treatment. Advanced patients have shorter survival than other subtypes. Maintenance therapy after combination chemotherapy can prolong the disease control time in patients with advanced TNBC. How to prolong the disease control time of patients with advanced TNBC without affecting the quality of life has become the focus of current research.

Anti-angiogenic drugs are currently one of the few targeted therapies that have achieved some efficacy in TNBC. Apatinib, a targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with breast cancer. The results of this study will help explore the new treatment of small molecule anti-angiogenic drugs for TNBC maintenance therapy, and provide some new ideas for improving individualized treatment options for patients with advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~75 years;
2. Triple-negative breast cancer (TNBC) confirmed by histology examination;
3. patients had received first-line combination chemotherapy for advanced metastatic disease, and had a complete response, partial response or stable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria;
4. received endocrine therapy for metastatic disease before first-line chemotherapy were allowed;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. A life expectancy of more than 12 weeks;
7. Baseline blood routine examination in accordance with the following criteria : ANC≥1.5×109/L，PLT≥90×109/L，Hb≥90g/L;
8. Liver and renal function in accordance with the following criteria: total bilirubin less than 1.5 times the upper limit of normal value; aspartate aminotransferase (AST), or alanine aminotransferase (ALT) less than 2.5 times the upper limit of normal value, less than 5 times the upper limit of normal value in patients with liver metastases.

   the creatinine clearance rate calculated greater than 60 mL/min;
9. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative, and they are willing to take effective contraceptive methods During the trial and within 8 weeks after the last dose;
10. Obtain informed consent from patients before starting any research-related operations and treatments to confirm that patients are willing to participate in this study and comply with research-related requirements.

Exclusion Criteria:

1. Metastasis/recurrence occurs within 6 months of adjuvant chemotherapy;
2. controlled high blood pressure, systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg;
3. urine routine test with urinary protein more than ++, or 24 hour urinary protein more than 1.0 g;
4. abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds or APTT >1.5 times the ULN);
5. Pregnant or lactating woman;
6. Symptomatic brain parenchymal and/or pia mater metastases without treatment and control;
7. Patients with Other malignant tumors in the past 5 years, except for fully treated cervical carcinoma in situ, cutaneous squamous cell carcinoma or well-controlled localized basal cell skin cancer;
8. Mental illness or other condition that affects patient compliance;
9. serious and uncontrollable systemic diseases (eg clinically significant cardiovascular disease, lung or metabolic disease, arteriovenous thrombosis, etc.) happened recently;
10. Can not take or absorb oral drugs;
11. Receiving any other testing drugs, or participating in other clinical trial 30 days before being enrolled in this trial;
12. The patient has previously received treatment with an anti-angiogenic drug (whether adjuvant or palliative);
13. Known or suspected to be allergic to any research drug or excipient;
14. Any other researcher believes that it is not appropriate to participate in this test.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-18 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | up to 6 months
  Time from randomization to disease progression or death for any cause

SECONDARY OUTCOMES:
overall survival | up to 6 months
  Time from randomization to death for any cause
tine to progress | up to 6 months
  Time from randomization to disease progression
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No